CLINICAL TRIAL: NCT07305142
Title: A Prospective, Randomized Controlled Study Comparing the Integrated Posterior-Anterior-Lateral (PAL) Approach and the Posterior Approach in Robot-Assisted Radical Prostatectomy: Evaluation of Perioperative Outcomes, Postoperative Functional Recovery, and Oncologic Control
Brief Title: Comparison of the Integrated Posterior-Anterior-Lateral Approach and the Posterior Approach in Robotic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xuepei Zhang, Director of Urology, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-KY-0820-002
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Urologic Cancer; Prostate; Robot Assisted Laparoscopic Radical Prostatectomy
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAL-RAPA (Active Comparator): Participants undergo robot-assisted laparoscopic radical prostatectomy(RAPA) via an integrated Posterior-Anterior-Lateral (PAL) approach using the da Vinci system.
  * Posterior:** mobilize sigmoid colon, incise rectovesical peritoneum, dissect vas deferens and seminal vesicles, open Denonvilliers' fascia, create a fascial window at prostate base.
  * Anterior:** enter retropubic space, preserve endopelvic fascia, puboprostatic ligaments, dorsal venous complex, expose bladder neck and anterior prostate.
  * Lateral:** dissect lateral bladder neck/prostate base, expand triangular space, retract seminal vesicle through posterior window, incise bladder neck, control vascular pedicles, perform atraumatic neurovascular bundle dissection, preserve urethral length.
  * Prostate removal** is followed by **continuous urethrovesical anastomosis** with 3-0 barbed suture.
  **Intended Purpose of Intervention:** Assess perioperative outcomes, early functional recovery, and oncologic safety of PAL-RAPA
  Interventions: Procedure: PAL combined approach group
- Posterior RAPA (Active Comparator): Participants undergo robot-assisted laparoscopic radical prostatectomy via a posterior-only approach using the da Vinci system. The procedure includes: mobilization of the sigmoid colon, incision of the rectovesical peritoneum, dissection of vas deferens and seminal vesicles, opening of Denonvilliers' fascia, and creation of a fascial window at the prostate base. Prostate removal is followed by continuous urethrovesical anastomosis using a 3-0 barbed suture.
  Interventions: Procedure: posterior approach group

INTERVENTIONS:
Procedure: PAL combined approach group — PAL combined approach was performed to resect the prostate
  Arms: PAL-RAPA
Procedure: posterior approach group — Intraoperative resection of the prostate was performed by posterior approach
  Arms: Posterior RAPA

SUMMARY:
This study aims to compare perioperative, pathological, and early functional outcomes of PAL （Posterior, Anterior and Lateral）combined approach RARP and posterior approach (with Retzius space preserved) RARP in the treatment of prostate cancer.The main question it aims to answer was:

What is the early therapeutic efficacy of robot-assisted laparoscopic radical prostatectomy using the combined posterior, anterior, and lateral (PAL) approach, and how does it compare with the traditional posterior approach? Participants were randomly assigned to undergo either robot-assisted laparoscopic radical prostatectomy using the PAL (posterior-anterior-lateral) approach or the classic posterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Prostate biopsy confirms prostate cancer;
* Clinical T stage <=T3a stage;
* Fully understand clinical trial protocols and sign informed consent;

Exclusion Criteria:

* Urinary incontinence before surgery;
* Previous endoscopic prostate surgery;
* There are serious underlying diseases that cannot tolerate surgery or have a survival of less than 5 years;
* Metastatic disease is present or lymph node involvement is suspected at diagnosis;
* Patients judged by the investigator to be unsuitable for participation in this clinical trial;

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
urinary continence | Patients were assessed for urinary incontinence, defined according to established criteria, via telephone at five time points after the removal of the urinary catheter (which was 2-3 weeks post-surgery): within 7 days, and at 1, 3, 6, and 12 months.
  was defined as the use of zero to one safety pad per day without any involuntary leakage.Immediate continence was defined as continence within seven days after catheter removal, while early continence was defined as continence achieved within three months.

SECONDARY OUTCOMES:
Operation time | During operation
Estimated blood loss | During operation
Complications | Perioperative
  Complications were classified according to the Clavien-Dindo system, and those of grade II or higher were documented in this study.
Time for removal of drainage tube | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: One year after the completion of the research

DOCUMENTS (2):
  • Study Protocol (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT07305142/Prot_000.pdf
  • Informed Consent Form (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT07305142/ICF_001.pdf